CLINICAL TRIAL: NCT00978848
Title: Non-Invasive Sexually Transmitted Disease Testing in Women Seeking Emergency Contraception or Urine Pregnancy Testing: Meeting the Needs of an At-Risk Population
Brief Title: Non-Invasive Sexually Transmitted Disease Testing in Women Seeking Emergency Contraception or Urine Pregnancy Testing
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Gen-Probe, Incorporated (Industry)
Responsible Party: Principal Investigator, Harold Wiesenfeld, Director, Division of Gynecologic Specialties & Division of Reproductive Infectious Diseases and Immunology, University of Pittsburgh
Other Study IDs: PRO8120077
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Trichomonas Vaginitis; Chlamydia Trachomatis; Neisseria Gonorrhoeae Infection
Keywords: trichomonas; chlamydia; gonorrhea; emergency contraception; emergency contraception use
MeSH Terms: conditions — Trichomonas Vaginitis; Gonorrhea; Trichomonas Infections; Chlamydia Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Any left over urine may be frozen for future use on infections in women
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women seeking emergency contraception: Women seeking emergency contraception
- Women seeking urine pregnancy testing: Women seeking urine pregnancy testing

SUMMARY:
The purpose of this study is to determine the prevalence and treatment rates of T. vaginalis, C. trachomatis, and N. gonorrhoeae in women seeking emergency contraception or urine pregnancy testing in the Magee-Womens Hospital outpatient clinic using a non-invasive urine STD test.

DETAILED DESCRIPTION:
This study has three primary objectives: 1) to determine the prevalence of T. vaginalis, C. trachomatis, and N. gonorrhoeae in women seeking emergency contraception or urine pregnancy testing - a population likely at increased risk of acquiring STDs; 2) to determine the rate of successful treatment in women diagnosed with STDs in this venue.

ELIGIBILITY:
Inclusion Criteria:

* Females at least age 15 at time of enrollment who are presenting at Magee-Womens Hospital for emergency contraception or urine pregnancy testing.
* Ability to provide written informed consent.

Exclusion Criteria:

* Diagnosis and/or treatment for an STD within 4 weeks of enrollment in the study.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Females at least age 15 at time of enrollment who are presenting at Magee-Womens Hospital for emergency contraception or urine pregnancy testing
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold C Wiesenfeld, MD, CM, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No